CLINICAL TRIAL: NCT05027360
Title: Sodium NItroPrusside Treatment in Acute Heart Failure: Multicenter, Observational, Retrospective Study
Brief Title: Sodium NItroPrusside Treatment in Acute Heart Failure
Acronym: SNIP-AHF
Status: Completed | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S_04_06_21_5186
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Acute Heart Failure
Keywords: Acute Heart Failure; sodium nitroprusside; NTproBNP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute heart Failure AHF: AHF diagnosis, defined as rapid onset or worsening of symptoms and/or signs of HF
  Interventions: Drug: SNP - Sodium Nitroprusside

INTERVENTIONS:
Drug: SNP - Sodium Nitroprusside — The primary objective of our study is to assess the efficacy and safety of SNP as part of the treatment regimen of AHF patients and to identify predictors of efficacy.

SUMMARY:
The primary objective of this multicentric observational retrospective study is to assess the efficacy and safety of SNP as part of the treatment regimen of AHF patients and to identify predictors of efficacy. The primary efficacy endpoint is brain natriuretic peptide (BNP) or N-terminal pro b-type natriuretic peptide (NT-proBNP) reduction (at least 25% from baseline levels) 48 hours after initiation of SNP infusion. AHF presentation (de novo or ADHF), systolic blood pression at presentation, left ventricle ejection fraction and dimension, entity of mitral regurgitation and central venous pressure will be evaluated in order to identify predictors of efficacy of SNP (in terms of primary endpoint).

DETAILED DESCRIPTION:
The present is a multicenter, observational, retrospective study. All consecutive patients admitted with a diagnosis of AHF to the Cardiothoracovascular Departments of the ASST Grande Ospedale Metropolitano Niguarda (Milan), ASST Ospedale Papa Giovanni XXIII (Bergamo) and Ospedale Le Molinette (Torino), and treated with intravenous SNP between January 2016 and January 2020 will be included, and medical records screened. Through the collaboration of the two joining institution, the investigator plan to include approximately 300 patients. Inclusion criteria are: age 18 years or older; AHF diagnosis, defined as rapid onset or worsening of symptoms and/or signs of HF; Intravenous SNP treatment. Exclusion criteria are: Age <18 years old; AHF after cardiac surgery; AHF complicated by cardiogenic shock requiring high dosage (defined as inotropic score >10) vasoactive agents and/or short-term extracorporeal life support (i.e. VA-ECMO, Impella). Inotropic score (IS) calculated as: dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 100 × norepinephrine dose (μg/kg/min) + 10 × phosphodiesterase 3 inhibitor dose (μg/kg/min). Invasive monitoring of central venous pressure (CVP) and arterial pressure may be present. The Swan Ganz pulmonary artery catheter for continuous haemodynamic monitoring will be rarely used. Simultaneous intravenous diuretics and concomitant inotropic agents with a maximun IS<20 administration will be tolerated. SNP will be administered intravenously by a continuous infusion at a dose of 0.2 up to 2 mcg/kg/min. Titration of SNP up to the maximum tolerated dose will be based on achieving decongestion, defined as decrease in CVP and reduction of pulmonary congestion, with a target mean arterial pressure of 65 to 70 mmHg. Headache or severe hypotension, as well as documented thiocyanate toxicity, will warrant discontinuation of SNP therapy. The primary objective of our study is to assess the efficacy and safety of SNP as part of the treatment regimen of AHF patients and to identify predictors of efficacy. The primary efficacy endpoint is brain natriuretic peptide (BNP) or N-terminal pro b-type natriuretic peptide (NT-proBNP) reduction (at least 25% from baseline levels) 48 hours after initiation of SNP infusion. Secondary endpoints include: Survival free from rehospitalization for HF at 6 months; 30-day and 6-month mortality; Composite of long-term LVAD implantation or HTx at 30 days and 6 months; Length of intensive care unit and total hospital stay. Safety endpoints are: thiocyanate toxicity, headache, severe hypotension requiring discontinuation of therapy, ventricular arrhythmias The investigators will evaluate the following baseline patients' characteristics in order to identify predictors of efficacy of SNP (in terms of primary endpoint): AHF presentation (de novo or ADHF); SBP at presentation (preserved, i.e. 90-140 mmHg; elevated, i.e. >140 mmHg; low, <90 mmHg); left ventricle ejection fraction (LVEF), graded as reduced (<40%), mid-range (40-49%) or preserved (≥50%); end-diastolic diameter (EDD); entity of mitral regurgitation (none/mild or moderate/severe mitral regurgitation); CVP (< 8 mmHg or ≥8 mmHg) Patient demographics, haemodynamics, laboratory values, echocardiographic parameters, adverse events and clinical outcomes will be obtained by complete chart review.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* AHF diagnosis, defined as rapid onset or worsening of symptoms and/or signs of HF. According to a recently proposed new definition, HF is a clinical syndrome with current or prior Symptoms and or signs caused by a structural and/or functional cardiac abnormality (as determined by EF <50%, abnormal cardiac chamber enlargement, E/E' >15, moderate/severe ventricular hypertrophy or moderate/severe valvular obstructive or regurgitant lesion) and corroborated by at least one of the following: Elevated natriuretic peptide levels ; Objective evidence of cardiogenic pulmonary or systemic congestion by diagnostic modalities such as imaging (e.g. by chest X-ray or elevated filling pressures by echocardiography) or haemodynamic measurement (e.g. right heart catheterization, pulmonary artery catheter) at rest or with provocation (e.g. exercise).
* Intravenous SNP treatment

Exclusion Criteria:

* Age <18 years old
* AHF after cardiac surgery
* AHF complicated by cardiogenic shock requiring high dosage (defined as inotropic score >10) vasoactive agents and/or short-term extracorporeal life support (i.e. VA-ECMO, Impella). Inotropic score (IS) calculated as: dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 100 × norepinephrine dose (μg/kg/min) + 10 × phosphodiesterase 3 inhibitor dose (μg/kg/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted with a diagnosis of AHF to the Cardiothoracovascular Departments of the ASST Grande Ospedale Metropolitano Niguarda (Milan), ASST Ospedale Papa Giovanni XXIII (Bergamo) and Ospedale Le Molinette (Torino), and treated with intravenous SNP between January 2016 and January 2020 will be included, and medical records screened. Through the collaboration of the two joining institution, we plan to include approximately 300 patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
NT-pro-BNP or BNP reduction | 48 hours
  Significant reduction (at least 25% from baseline levels) 48 hours after initiation of SNP infusion

SECONDARY OUTCOMES:
Hospitalizations | 6 months
  Survival free from re-hospitalizations for heart failure
Mortality | 30 days and 6 months
  All-cause mortality
Heart replacement therapies | 30 days and 6 months
  Composite of long-term LVAD implantation or HTx
Intensive Care Unit | through study completion, an average of 6 months
  Length of intensive care unit and total hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided

REFERENCES:
- [Derived] Garatti L, Frea S, Bocchino PP, Angelini F, Cingolani M, Sacco A, Rondinara GM, Bagnardi V, Sala IM, Kapur NK, Colombo PC, De Ferrari GM, Morici N. Sodium nitroprusside in acute heart failure: A multicenter historic cohort study. Int J Cardiol. 2022 Dec 15;369:37-44. doi: 10.1016/j.ijcard.2022.08.009. Epub 2022 Aug 6. PMID 35944767